CLINICAL TRIAL: NCT04794374
Title: Effects of Telerehabilitation After Discharge on Quality of Life, Psychosocial Status, Physical Activity, Daily Activities of Living, and Sleep Quality in Patients Treated as Inpatients With the Diagnosis of COVID-19
Brief Title: Effects of Telerehabilitation After Discharge in COVID-19 Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aslihan Cakmak, Principal Investigator, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KA-20085
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Covid19
Keywords: telerehabilitation; physical activity; sleep quality; post COVID-19; quality of life
MeSH Terms: conditions — COVID-19; Motor Activity; Sleep Initiation and Maintenance Disorders | interventions — Telerehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Discharged COVID-19 survivors (Experimental): Telerehabilitation will be provided by physiotherapists including audio, video visits.
  A brochure designed by physiotherapists for COVID-19 survivors will be used. Physiotherapists will call patients weekly and guide, design, modify the exercises accordingly to the patients.
  Interventions: Other: Telerehabilitation

INTERVENTIONS:
Other: Telerehabilitation — Telerehabilitation will consists of physiotherapist-guided exercises. Exercises will be designed by physiotherapists for COVID-19 survivors using the current guidelines. Exercise brochure will be prepared and will be sent to participants. Repetitions and sets of exercises will be modified according to the patients.

SUMMARY:
Effects of telerehabilitation after discharge on quality of Life, psychosocial status, physical activity, daily activities of living, and sleep quality in patients treated as inpatients with the diagnosis of COVID-19 will be investigated. Post-discharge physical activity level, psychosocial status, sleep quality, quality of life, daily activities of living, and quality of life will be determined. The effects of exercise interventions in online-based physiotherapist monitoring will be provided. Monthly comparisons of physical activity, quality of life, depression, and sleep quality responses using telerehabilitation for three months following COVID-19 will be investigated.

DETAILED DESCRIPTION:
The new type of Coronavirus (SARS-CoV-2) has progressed rapidly in our country and around the world and has caused a global health emergency, requiring the implementation of restrictive measures. While the origin of SARS-CoV-2 is still under investigation, the available information points to wild animals sold illegally in the Wuhan Seafood Wholesale Market. Common symptoms of infection are fever, cough, and dyspnea. In more severe cases, pneumonia, severe acute respiratory tract infection, renal failure, and even death may occur. Up-to-date information about physiotherapy and rehabilitation applications on COVID-19 disease is limited to positioning and mobilization in the acute phase of the disease. Current guidelines and protocols state that airway clearance techniques, respiratory exercises and practices using assistive devices, exercise training and respiratory muscle training should not be applied in the acute period. Tele-medicine is a clinical practice that connects the patient to healthcare professionals through electronic platforms, potentially improving the self-management of patients and allowing the care of patients with limited access to health services. In these days when staying at home is recommended to minimize exposure and contamination risk, telerehabilitation can be considered as an advantage, using information and communication technologies to provide remote rehabilitation services to individuals at home. It has been reported that with telerehabilitation, improvements have been achieved in health outcomes and quality of life, such as reducing hospitalization rates and re-admissions, ensuring early discharge, facilitating access to rehabilitation services, decreasing costs, and ensuring early return to work. Regular physical activity and exercise provide many health benefits, such as increasing cardiorespiratory fitness and reducing symptoms of anxiety and depression. Increasing cardiorespiratory fitness may play a preventive and facilitating role against respiratory infections. This may prevent or help treat pneumonia and acute respiratory distress syndrome, which develops with COVID-19 and causes respiratory failure. It has been stated that there is a significant decrease in the level of physical activity globally in the period of social isolation, which is accepted worldwide during COVID-19 pandemic. Decrease in the level of physical activity and increase in sedentary behavior due to isolation limitations may cause rapid deterioration and premature death in cardiovascular health in a population with high cardiovascular risk. Considering that short-term (1-4 weeks) inactivity is associated with adverse effects on cardiovascular function and structure, and increased cardiovascular risk factors, it appears to be a clinically relevant intervention to promote the health benefits of home-based physical activity programs. In this study, a brochure created by physiotherapists for post-COVID-19 patients will be sent electronically. The number of repetitions and/or sets of the exercises in the brochure will be increased weekly by the physiotherapists according to the tolerance of the patients. Physical activity levels will be questioned at the beginning and at the end of each month to be maintained for three months in total. The need for isolation due to the COVID-19 pandemic creates an unprecedented, stressful situation for many people for an unknown period of time. In addition to increasing the level of anxiety and depression, this may have negative effects on sleep quality. Since sleep plays a main role in emotion regulation, sleep disturbances may have direct consequences on emotional functioning. Therefore, it was planned to evaluate depression and sleep in individuals who survived COVID-19 at the beginning and at the end of each month, for a total of three months. It will be possible to determine whether there is a relationship between depression and sleep efficiency with exercise recommendations that will be given in a controlled manner by a physiotherapist via telerehabilitation and increase according to the patient's tolerance. It has been reported that patients hospitalized with acute respiratory distress syndrome have post-traumatic stress disorder at a rate of 22% -24%, depression at a rate of 26% -33%, and general anxiety at a rate of 38% -44% even after 2 years. It has been reported that these are concerns that may accompany a serious decrease in quality of life and function after COVID-19. Therefore, it is planned to assess quality of life at the beginning and at the end of each month for a total of three months in individuals who survived COVID-19.

Post-discharge physical activity level, psychosocial status, sleep quality, quality of life, daily activities of living, and quality of life will be determined. The effect of exercise interventions in online-based physiotherapist monitoring will be provided. Monthly comparisons of physical activity, quality of life, depression, and sleep quality responses using telerehabilitation for three months following COVID-19 will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Being clinically stable,
* Being 18 years old or older
* Being a volunteer for the study and providing their consent,
* Able to read and write
* Having a smart phone and being able to use it

Exclusion Criteria:

* Having unstable clinical condition
* Having severe neuromuscular and musculoskeletal problems,
* Being unable to cooperate and respond to the questionnaires and scales
* Not being a volunteer to participate

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2021-10-27 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Physical activity level | up to 6 months
  Turkish version of the International Physical Activity Questionnaire (IPAQ) short form will be used for the assessment of physical activity. The IPAQ short form is a questionnaire consisting of seven questions used to evaluate the level of physical activity in people aged 18-69 years. Walking, moderate activity duration, and vigorous activity duration are the sub-parameters of the questionnaire. The sitting time is evaluated separately. The total score of the questionnaire is obtained by the sum of the products of metabolic equivalent (MET), activity duration (minutes) and frequency (days) corresponding to the activity. The questionnaire has Turkish validity and reliability.
Psychosocial status | up to 6 months
  Psychosocial status will be evaluated using the Turkish version of Hospital Anxiety and Depression Scale (HADS). HADS will be used to assess the level of anxiety and depression. This scale is a 14-item self-report scale that aims to determine the risk in terms of anxiety and depression in the patient, and measure its level and change in severity. The scale, which was asked to be answered considering the last few days, has two subscales, consisting of seven items measuring anxiety and seven items measuring depression. Higher scores indicate better psychosocial status.
Sleep quality | up to 6 months
  Evaluation of sleep quality will be assessed using Pittsburgh Sleep Quality Index (PSQI). PSQI is a self-report scale that evaluates sleep quality and sleep disturbance over a one-month period. PSQI includes seven components and 19 questions. The components include perceived sleep quality, sleep delay (how long it takes to fall asleep), sleep time, habitual sleep activity (how much a person is asleep compared to the time spent in bed), sleep disturbances (noise, temperature, pain, nocturia), sleep medications, and daytime dysfunction (drowsiness, concentration). The total score ranges from 0 to 21. A score higher than five indicates sleep disorder. The Turkish validity and reliability study of this questionnaire was conducted.
Health related quality of life | up to 6 months
  Nottingham Health Profile (NHP) will be used to assess quality of life. This questionnaire is a general quality of life scale developed to measure perceived health problems and the extent to which these problems affect normal daily activities. The scale assesses the perceived restriction or discomfort in 6 sub-sections: energy (3 items), pain (8 items), emotional reactions (9 items), sleep (5 items), social isolation (5 items), and physical activity (8 items). There are 38 items. There is a possible score limit ranging from 0-100 for each subsection. "0 points" indicates that there is no restriction. "100 points" indicates the presence of all restrictions listed. There is a Turkish validity and reliability study of the NHP.
Activities of daily living | up to 6 months
  The Barthel Index basically evaluates mobility and self-care activities. It consists of 10 sub-headings: eating, bathing, self-care, dressing, bladder control, bowel control, toilet use, chair / bed transfer, mobility, and use of stairs. The total score ranges from 0 to 100. "0" points total addiction; A score of "100" indicates complete independence. The Barthel Index has Turkish validity and reliability.

CONTACTS AND LOCATIONS:
Overall Officials: Lale Ozisik, Assoc.Prof., Study Chair — Hacettepe University; Nursel Calik Basaran, Asst.Prof, Study Chair — Hacettepe University; Oguz Abdullah Uyaroglu, Asst.Prof, Principal Investigator — Hacettepe University; Deniz Inal-Ince, Prof., Study Chair — Hacettepe University; Naciye Vardar-Yagli, Assoc.Prof., Study Chair — Hacettepe University; Melda Saglam, Assoc.Prof., Study Chair — Hacettepe University; Ebru Calik-Kutukcu, Assoc.Prof., Principal Investigator — Hacettepe University; Esra Kinaci, MSc, PT., Principal Investigator — Hacettepe University; Gulay Sain Guven, Prof., Study Director — Hacettepe University; Aslihan Cakmak, MSc, PT., Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] COVID-19 (SARS-CoV2) Enfeksiyonu Rehberi (Bilim Kurulu Çalışması). T.C. Sağlık Bakanlığı. Halk Sağlığı Genel Müdürlüğü. T.C. Sağlık Bakanlığı. (https://covid19bilgi.saglik.gov.tr/depo/rehberler/COVID-19_Rehberi.pdf) Erişim Tarihi: 19 Mayıs 2020.
- [Background] Mohamed AA, Alawna M. Role of increasing the aerobic capacity on improving the function of immune and respiratory systems in patients with coronavirus (COVID-19): A review. Diabetes Metab Syndr. 2020 Jul-Aug;14(4):489-496. doi: 10.1016/j.dsx.2020.04.038. Epub 2020 Apr 28. PMID 32388326
- [Background] İnal İnce D, Vardar Yağlı N, Sağlam M, Çalık Kütükcü E. COVID-19 Enfeksiyonunda Akut ve Post-Akut Fizyoterapi ve Rehabilitasyon. Turk J Physiother Rehabil. 2020;31(1):81-93.
- [Background] Ambrosino N, Fracchia C. The role of tele-medicine in patients with respiratory diseases. Expert Rev Respir Med. 2017 Nov;11(11):893-900. doi: 10.1080/17476348.2017.1383898. Epub 2017 Sep 27. PMID 28942692
- [Background] Galea MD. Telemedicine in Rehabilitation. Phys Med Rehabil Clin N Am. 2019 May;30(2):473-483. doi: 10.1016/j.pmr.2018.12.002. Epub 2019 Mar 5. PMID 30954160
- [Background] Global Recommendations on Physical Activity for Health. Geneva: World Health Organization; 2010. Available from http://www.ncbi.nlm.nih.gov/books/NBK305057/ PMID 26180873
- [Background] Pecanha T, Goessler KF, Roschel H, Gualano B. Social isolation during the COVID-19 pandemic can increase physical inactivity and the global burden of cardiovascular disease. Am J Physiol Heart Circ Physiol. 2020 Jun 1;318(6):H1441-H1446. doi: 10.1152/ajpheart.00268.2020. Epub 2020 May 15. PMID 32412779
- [Background] Altena E, Baglioni C, Espie CA, Ellis J, Gavriloff D, Holzinger B, Schlarb A, Frase L, Jernelov S, Riemann D. Dealing with sleep problems during home confinement due to the COVID-19 outbreak: Practical recommendations from a task force of the European CBT-I Academy. J Sleep Res. 2020 Aug;29(4):e13052. doi: 10.1111/jsr.13052. Epub 2020 May 4. PMID 32246787
- [Background] Herridge MS, Moss M, Hough CL, Hopkins RO, Rice TW, Bienvenu OJ, Azoulay E. Recovery and outcomes after the acute respiratory distress syndrome (ARDS) in patients and their family caregivers. Intensive Care Med. 2016 May;42(5):725-738. doi: 10.1007/s00134-016-4321-8. Epub 2016 Mar 30. PMID 27025938
- [Background] Sheehy LM. Considerations for Postacute Rehabilitation for Survivors of COVID-19. JMIR Public Health Surveill. 2020 May 8;6(2):e19462. doi: 10.2196/19462. PMID 32369030
- [Background] Vitacca M, Carone M, Clini EM, Paneroni M, Lazzeri M, Lanza A, Privitera E, Pasqua F, Gigliotti F, Castellana G, Banfi P, Guffanti E, Santus P, Ambrosino N; ITS - AIPO, the ARIR and the SIP/IRS. Joint Statement on the Role of Respiratory Rehabilitation in the COVID-19 Crisis: The Italian Position Paper. Respiration. 2020;99(6):493-499. doi: 10.1159/000508399. Epub 2020 May 19. PMID 32428909
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Saglam M, Arikan H, Savci S, Inal-Ince D, Bosnak-Guclu M, Karabulut E, Tokgozoglu L. International physical activity questionnaire: reliability and validity of the Turkish version. Percept Mot Skills. 2010 Aug;111(1):278-84. doi: 10.2466/06.08.PMS.111.4.278-284. PMID 21058606
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Aydemir Ö, Güvenir T, Küey L, Kültür S. Hastane Anksiyete ve Depresyon Ölçeği Türkçe Formunun Geçerlilik ve Güvenilirlik Çalışması Türk Psikiyatri Derg. 1997;8(4):280-7.
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Ağargün MY, Kara H, Anlar Ö. Pittsburgh Uyku Kalite İndeksinin Geçerliği ve Güvenirliği. Türk Psikiyatri Derg. 1996;7(2):107-15.
- [Background] Hunt SM, McKenna SP, McEwen J, Backett EM, Williams J, Papp E. A quantitative approach to perceived health status: a validation study. J Epidemiol Community Health. 1980 Dec;34(4):281-6. doi: 10.1136/jech.34.4.281. PMID 7241028
- [Background] Kucukdeveci AA, McKenna SP, Kutlay S, Gursel Y, Whalley D, Arasil T. The development and psychometric assessment of the Turkish version of the Nottingham Health Profile. Int J Rehabil Res. 2000 Mar;23(1):31-8. doi: 10.1097/00004356-200023010-00004. PMID 10826123
- [Background] MAHONEY FI, BARTHEL DW. FUNCTIONAL EVALUATION: THE BARTHEL INDEX. Md State Med J. 1965 Feb;14:61-5. No abstract available. PMID 14258950
- [Background] Kucukdeveci AA, Yavuzer G, Tennant A, Suldur N, Sonel B, Arasil T. Adaptation of the modified Barthel Index for use in physical medicine and rehabilitation in Turkey. Scand J Rehabil Med. 2000 Jun;32(2):87-92. PMID 10853723